CLINICAL TRIAL: NCT06245876
Title: Lung EpiCheck Biomarkers Development Study
Status: Recruiting | Type: Observational
Sponsor: Nucleix Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Evergreen-LNG-001
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Lung Cancer
Keywords: Lung cancer screening
MeSH Terms: conditions — Lung Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cases Cohort: Subjects age 50-80 years old, with smoking history of at least 20 pack years with either (a) a high suspicion for lung cancer, who are planned to undergo biopsy or surgery to establish a definitive diagnosis after enrollment; or (b) confirmed primary lung cancer diagnosis, treatment naïve subjects.
  Interventions: Other: Blood collection
- USPSTF At Risk - Control Cohort: Healthy subjects aged 50-80 years old with smoking history of at least 20 pack years.
  Interventions: Other: Blood collection
- Healthy Control Cohort: Healthy subjects aged 20-80 years old which are non-smokers or with smoking history of less than 20 pack years.
  Interventions: Other: Blood collection

INTERVENTIONS:
Other: Blood collection — Blood collection

SUMMARY:
This study is part of the development of a non-invasive lung cancer screening test which aim to identify early-stage lung cancer in patients at high risk for lung cancer.

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational nonsignificant risk study aimed to collect blood and clinical data from primary lung cancer and control subjects to characterize various biomarkers that will discriminate between lung cancer and control subjects.

ELIGIBILITY:
Inclusion Criteria - Cases:

* Age 50-80 years
* Subjects who are currently smoking or former smokers, with at least 20 pack-years
* Subjects with either A high suspicion for lung cancer, with planned biopsy or surgery to establish a definitive diagnosis within 60 days after enrollment or treatment naive lung cancer patients confirmed by pathology.

Exclusion Criteria - Cases

* Known diagnosis or treatment of cancer from any kind in the past 5 years, except of fully resected non-melanoma skin cancer or fully-resected carcinoma in situ of the cervix and except from the current lung cancer

Inclusion Criteria - USPSTF risk

* Age 50-80 years
* Subjects who are currently smoking or former smokers, with at least 20 pack-years

Exclusion Criteria - USPSTF risk

- Known diagnosis or treatment of cancer of any kind in the past 5 years, except for fully resected non-melanoma skin cancer or fully-resected carcinoma in situ of the cervix

Inclusion Criteria - Healthy controls

* Age 20-80 years
* Never smoker or current / previous smoker < 20 pack year history

Exclusion Criteria - Healthy Controls

* Known diagnosis or treatment of cancer of any kind in the past (lifetime), except for fully resected non-melanoma skin cancer or fully-resected carcinoma in situ of the cervix.
* Not previously diagnosed with a lung lesion highly suspicious for cancer
* Under follow up or work up for any lesion suspicious for any type of cancer
* Presenting with fever with body temperature 100.4°F (38°C) or higher
* Acute exacerbation or flare of an inflammatory condition requiring escalation in medical therapy within 14 days prior to blood draw
* Pregnancy
* Any history of blood product transfusion within 30 days prior to blood draw

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects should be without other cancer in the past 5 years except for fully resected non-melanoma skin cancer or fully-resected carcinoma in situ of the cervix
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Performance | Day 1
  Performance of the assay in terms of (1) Sensitivity (2) Specificity (3) NPV (negative predictive value) and (4) PPV (positive predictive value).

CONTACTS AND LOCATIONS:
Locations (10):
- United States (6):
  - Life Spring Clinical Research, Miami, Florida
  - Emerald Coast OBGYN, Panama City, Florida
  - Ochsner LSU Health Shreveport - Regional Urology, Shreveport, Louisiana
  - Comprehensive Urology, Southfield, Michigan
  - Michigan Institute of Urology, P.C., Troy, Michigan
  - Urology San Antonio, San Antonio, Texas
- National Koranyi Institute for Pulmonology, Budapest, Hungary
- Israel (2):
  - Carmel Medical Center, Haifa
  - Sourasky Medical Center, Tel Aviv
- ZGT Medical Center, Hengelo, Netherlands

IPD SHARING:
Plan to Share IPD: No